CLINICAL TRIAL: NCT04167826
Title: Oral Health Status and Diet History Analysis Among Orphan House Children From 10-14 Years in Cairo Governorate : A Cross Sectional Study
Brief Title: Oral Health Status and Diet History Analysis Among Orphan House Children From 10-14 Years in Cairo Governorate.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulrahman mohamed salah, Master student in Cairo university, Cairo University
Other Study IDs: CEBD-CU-2019-11-14
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Gingival Disease Due to Bacteria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the purpose of study to determine oral health status and dietary habits among group of orphan children from 10-14 years in Cairo Governorate.

DETAILED DESCRIPTION:
The study's investigators will record all data related to oral health status of orphan children from 10-14 years and their dietary habits to describe usual food intake and its variation over a long period of time . the OHI-S will also recorded which has 2 components the Debris index and Calculus index .

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children aged from 10-14 years
* Cooperative children

Exclusion Criteria:

* Children with systemic disease , genetic disorders , or any disabilities

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will done for Orphan children in Resalaa charity organization in Cairo governorate in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
oral health status | 3 months
  Debris index
oral health status | 3 months
  Calculus index
Diet history analysis | 3 months
  Diet history chart

CONTACTS AND LOCATIONS:
Overall Officials: Sherine Ezz eldeen, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided